CLINICAL TRIAL: NCT05531474
Title: Bariatric Surgery for the Reduction of CArdioVascular Events Randomized Controlled Trial
Acronym: BRAVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRAVE-Full Trial
Record Dates: First submitted 2022-06-13; First posted 2022-09-08 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Complication; Bariatric Surgery Candidate
MeSH Terms: interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medical Weight Management (Active Comparator): MWM corresponds to standard medical practice for weight loss that is available at the local participating centre, and thus reflects the local standard of care. MWM will typically consist of dietary, lifestyle and/or behavioral modification counseling, which may include nutritional counseling, safe weight management and/or making healthy lifestyle changes. MWM may also include the implementation of a low caloric diet, which may comprise the use of adjuvant meal replacements and/or anti-obesity mediations at the discretion of the treating physician and according to local practice guidelines.
  Interventions: Behavioral: Medical Weight Management
- Bariatric Surgery (Experimental): The bariatric surgery procedures performed in BRAVE include either gastric bypass, sleeve gastrectomy, or duodenal switch, performed at the discretion of the surgeon and according to local practice standards. Sleeve gastrectomy will be performed as a stand-alone procedure, but may also be performed as part of a planned duodenal switch. Gastric banding is not permitted. Patients may receive a low fat, high protein meal replacement preceding surgery to reduce the size of the liver. Perioperative use of aspirin, thienopyridines (clopidogrel, ticagrelor or prasugrel), and anti-thrombotic therapy (compression stockings and subcutaneous heparin) should follow local guidelines and will be left at the discretion of the individual surgeons. .
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Procedure: Bariatric Surgery — Bariatric surgery involves either gastric bypass, sleeve gastrectomy, or duodenal switch, performed at the discretion of the surgeon and according to local practice standards.
  Arms: Bariatric Surgery
Behavioral: Medical Weight Management — The current standard medical practice for weight loss that is available at the local participating centre, reflecting the local standard of care
  Arms: Medical Weight Management

SUMMARY:
The primary objective of this study is to evaluate if, in patients with severe obesity (body mass index (BMI) ≥30 kg/m2) and high-risk cardiovascular disease (CVD), bariatric surgery compared to medical weight management (MWM) safely reduces the risk of major cardiovascular events. The cost-effectiveness of bariatric surgery will also be examined. Separate sub-studies will be performed to examine the relationship between bariatric surgery and mental health, cardiac structure and function, genomics, proteomics and metabolomics.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index ≥30 kg/m2; OR BMI ≥30 kg/m2 to 34.9 kg/m2 and have type 2 diabetes or are >55 years of age
2. Age ≥18 years
3. High-risk CVD, defined as the presence of any one of the following:

   1. High-risk coronary artery disease (CAD) (i.e., history of MI, percutaneous coronary intervention, coronary artery bypass grafting, or stenoses ≥ 50% in 2 or more major coronary arteries)
   2. Left ventricular ejection fraction (LVEF) < 40%
   3. Heart failure with preserved ejection fraction (LVEF > 40%) and either HF hospitalization in the last 2-years or N-terminal pro b-type natriuretic peptide (NT-proBNP) > 300 pg/ml or BNP > 100 pg/ml in the past 12 months
   4. Documented atrial fibrillation (AF) with CHA2DS2-VASc ≥2 stroke risk score
   5. History of any stroke
   6. Documented peripheral arterial disease (PAD) (i.e., peripheral revascularization of the iliac, infra-inguinal or carotid arteries; limb or foot amputation for arterial vascular disease; or ≥50% carotid or peripheral artery stenosis)

Exclusion Criteria:

1. Hospital admission for HF, myocardial infarction, stroke or coronary revascularization within 30 days of randomization
2. Percutaneous coronary intervention with a drug eluting stent within 90 days of randomization.
3. Pregnancy
4. Contraindication to bariatric surgery
5. Prior bariatric surgery, other than gastric banding
6. Life expectancy <2 years from non-cardiovascular causes
7. Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Outcomes | Through study completion, expected average of 6 years
  Composite of cardiovascular mortality, myocardial infarction (MI), stroke, and hospitalization for heart failure (HF).

SECONDARY OUTCOMES:
All-cause mortality | Through study completion, expected average of 6 years
Cardiovascular mortality | Through study completion, expected average of 6 years
Myocardial infarction | Through study completion, expected average of 6 years
Stroke | Through study completion, expected average of 6 years
Hospitalization for heart failure | Through study completion, expected average of 6 years
New onset or remission of type 2 diabetes as per Diabetes Canada / American Diabetes Association Guidelines | Through study completion, expected average of 6 years
New onset atrial fibrillation as assessed by ECG or heart rhythm monitoring | Through study completion, expected average of 6 years
Cost effectiveness analysis, measured in quality adjusted life years | Through study completion, expected average of 6 years
  Economic evaluation to compare the costs and health outcomes associated with bariatric surgery and medical weight management

OTHER OUTCOMES:
Change in quality of life assessed by EQ5D questionnaire | Through study completion, expected average of 6 years
Change in quality of life assessed by Laval questionnaire | Through study completion, expected average of 6 years
Change in weight | Through study completion, expected average of 6 years
Number of hospital admissions irrespective of cause | Through study completion, expected average of 6 years
Number of participants with a new cancer diagnosis | Through study completion, expected average of 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Salim Yusuf, DPhil, DSc (Oxon), FRCPC, FRSC, Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No